CLINICAL TRIAL: NCT03654573
Title: The MOCA I Study - Microvascular Obstruction with CoFI™ System Assessment
Acronym: MOCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CorFlow Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1801
Record Dates: First submitted 2018-08-16; First posted 2018-08-31 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Microvascular Obstruction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: N= 50 Diagnostic and N= 20 Therapeutic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STEMI patients (Experimental): Adult subjects presenting with STEMI in the LAD undergoing PPCI
  Interventions: Device: CorFlow Controlled Flow Infusion System - CoFI™

INTERVENTIONS:
Device: CorFlow Controlled Flow Infusion System - CoFI™ — The CorFlow CoFI™ System is intended to assess the dynamic microvascular resistance and to treat microvascular obstruction in the coronary vasculature of patients following PCI with stent placement.

SUMMARY:
First-in-Human study to assess the CoFI™ device related safety and the feasibility of the diagnostic and the therapeutic sequence as well as the correlation between the dynamic microvascular resistance (dMVR) and microvascular obstruction (MVO) as measured by MRI in patients presenting with acute ST-elevation myocardial infarction (STEMI) undergoing percutaneous coronary intervention (PCI).

ELIGIBILITY:
Major Inclusion Criteria:

* Patients 18 years of age or older presenting with ST-elevation myocardial infarction in the left anterior descending artery (LAD) undergoing primary percutaneous coronary intervention.
* Competent mental condition to provide signed and dated ethics committee approved study consent prior to study related procedures
* Eligible for prasugrel, ticagrelor, cangrelor, tirofiban, UFH and GP IIb/IIIa inhibitors
* Referred for primary PCI within 5 hours of symptom onset with evidence of continuing ischemia and symptom to balloon time not exceeding 6 hours

Major Exclusion Criteria:

* Unconsciousness
* Previous bypass graft surgery
* Contraindication to CMRI
* Recent or current major bleeding within 30 days prior to intervention
* Recent major surgery within 30 days prior to intervention
* End-stage heart failure with inotrope support and/or consideration for LVAD or heart transplant
* Transient ischemic attack or stroke within 30 days prior to intervention
* Pregnant or females of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
The incidence of study device or study procedure adverse effect or event | up to 30 days
  Safety Objective is the incidence of study device or study procedure adverse effect or event at up to 30 days. To assess the CoFI™ device related safety and the feasibility of the diagnostic and the therapeutic sequence as well as the correlation between the dynamic microvascular resistance (dMVR) and microvascular obstruction (MVO) as measured by MRI in patients presenting with acute ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI).

SECONDARY OUTCOMES:
Diagnostic Success | 0 days
  Ability to perform a diagnostic sequence and to calculate a base flow resistance curve
Therapeutic Success | 0 days
  Ability to perform the therapeutic sequence as described in the CIP

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hunziker, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (8):
- Lithuania (2):
  - The Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Switzerland (5):
  - Inselspital Bern, Bern, Canton of Bern
  - Cardiocentro Ticino, Lugano, Canton Ticino
  - HUG Geneva, Geneva
  - CHUV Lausanne, Lausanne
  - UniversitätsSpital Zürich, Zurich
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No